CLINICAL TRIAL: NCT01133938
Title: Predictive Factors for the Development of Osteonecrosis After the Treatment of the Developmental Dislocated Hip. A Comparison of Early Open Reduction Versus Late Open Reduction With Combined Pemberton and Femoral Osteotomies
Brief Title: Predictive Factors for the Development of Osteonecrosis After the Treatment of the Developmental Dislocated Hip
Status: Completed | Type: Observational
Sponsor: Orthopedic Hospital Vienna Speising (Other)
Responsible Party: Orthopedic Hospital Vienna Speising, Orthopedic Hospital Vienna Speising
Other Study IDs: OR-27052010
Record Dates: First submitted 2010-05-28; First posted 2010-05-31 (Estimated); Last update posted 2010-06-03 (Estimated); Status verified 2010-05

CONDITIONS: Predictors of Osteonecrosis of the Femoral Head After Treatment of the Dislocated Hip

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Closed reduction < 12 months of age
- Open reduction < 12 months of age
- Open reduction with concomitant osteotomies > 12 months fo age

SUMMARY:
Several risk factors for the development of osteonecrosis of the femoral head following treatment of developmental dislocated hip have been reported. The need for further research with a large-enough sample size including statistical adjustment of confounders was demanded. The purpose of the present study was to find reliable predictors of osteonecrosis in patients managed for developmental dislocation of the hip and to evaluate if delayed treatment increased the risk of residual acetabular dysplasia requiring secondary surgeries.

ELIGIBILITY:
Inclusion Criteria:

* Follow-up > 3 years

Exclusion Criteria:

* teratological hip dislocation
* neuromuscular disease
* previous open reduction at another medical institution

Ages: 1 Month to 15 Years | Sex: All
Age Groups: Child
Study Population: Consecutive series of patients hospitalized because of developmental dislocated hip between 1198 and February 2007
Sampling Method: Probability Sample
Enrollment: 79 (Actual)
Dates: Start 2009-01; Primary Completion 2010-02 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Osteonecrosis of the femoral head

SECONDARY OUTCOMES:
Secondary reconstructive procedures due to residual acetabular dysplasia

CONTACTS AND LOCATIONS:
Locations (1):
- Orthopedic Hospital Vienna Speising, Vienna, Vienna, Austria